CLINICAL TRIAL: NCT03714919
Title: A Pilot Study: a Non-opioid Technique for Postoperative Adenoidectomy Pain Relief in Pediatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arlyne Thung (Other)
Responsible Party: Sponsor-Investigator, Arlyne Thung, Attending Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-00235
Record Dates: First submitted 2018-10-19; First posted 2018-10-22 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Adenoid Hypertrophy
MeSH Terms: interventions — Dextromethorphan; Acetylcysteine; Acetaminophen; Dexmedetomidine; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Non-opiod pain relief (Experimental): Subjects will receive preoperative oral dextromethorphan & acetaminophen and intraoperative intravenous dexmedetomidine & ketamine.
  Interventions: Drug: Dextromethorphan; Drug: Acetaminophen; Drug: Dexmedetomidine; Drug: Ketamine

INTERVENTIONS:
Drug: Dextromethorphan — Preoperative oral dextromethorphan 1 mg/kg
  Other Names: Robitussin
Drug: Acetaminophen — Preoperative oral acetaminophen 15 mg/kg
  Other Names: Tylenol
Drug: Dexmedetomidine — Intraoperative intravenous dexmedetomidine 0.5 μg/kg
  Other Names: Precedex
Drug: Ketamine — Intraoperative intravenous ketamine 0.5 mg/kg
  Other Names: Ketalar

SUMMARY:
This proposed study will assess analgesic efficacy of a multi-modal, non-opioid analgesic regimen for providing surgical analgesia in pediatric patients undergoing adenoidectomy and to assess recovery characteristics in the post-anesthesia care unit (PACU) and at home following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing adenoidectomy ± bilateral ear tube placement
2. Have a parent/guardian who are compliant with routine medical care, capable of subjective evaluation and able to read, understand and sign the informed consent in accordance with IRB regulations

Exclusion Criteria:

1. An American Society of Anesthesiologists Physical Status ≥ 4 (severe disease that is life threatening);
2. A known hypersensitivity or allergy to any of the study medications;
3. A history of chronic opioid use prior to surgery;
4. Coexisting renal or hepatic disease;
5. Morbid obesity (BMI% ≥ 99).

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlyne Thung, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-opiod Pain Relief
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Non-opiod Pain Relief
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5 [3 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Weight [Median (Inter-Quartile Range); unit: kilograms] | 20.5 [16.65 to 25.175]
Height [Median (Inter-Quartile Range); unit: centimeters] | 110 [101.5 to 118.35]
ASA 1 [Number; unit: participants] — The American Society of Anesthesiologists (ASA) physical status classification 1 = normal healthy patient
  participants | 6
ASA 2 [Number; unit: participants] — The American Society of Anesthesiologists (ASA) physical status classification 2 = patient with mild systemic disease
  participants | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Score
Description: Visual Analogue Scale (VAS) pain scores (0 being no pain and 10 being worst pain) in post-anesthesia care unit (PACU).
Time Frame: 1 hr post-op
Measure: Mean (Standard Deviation); unit: pain score
Arm/Group | Non-opiod Pain Relief
Number analyzed (Participants) | 10
pain score | 0 (0)

2. Secondary Outcome: Extubation Time
Description: Amount of time in the PACU before patient is ready to be extubated.
Time Frame: 1 hr post-op
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Non-opiod Pain Relief
Number analyzed (Participants) | 10
minutes | 23 [17 to 29]

3. Secondary Outcome: Time in PACU
Description: Total time in PACU before patient met discharge criteria.
Time Frame: 1-2 hr post-op
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Non-opiod Pain Relief
Number analyzed (Participants) | 10
minutes | 56 [49 to 65]

4. Secondary Outcome: Number of Participants With Sedation, Nausea/Vomiting, or Hallucinations
Description: Presence of sedation, nausea/vomiting, or hallucinations post-operatively.
Time Frame: 2 hours post-op
Measure: Number; unit: participants
Arm/Group | Non-opiod Pain Relief
Number analyzed (Participants) | 10
participants
  Sedation | 7
  Nausea/Vomiting | 1
  Hallucinations | 0

5. Secondary Outcome: End of Surgery to Hospital Discharge
Description: Length of time before patient is ready to be discharged home.
Time Frame: 2-3 hours post-op
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Non-opiod Pain Relief
Number analyzed (Participants) | 10
minutes | 122 [106 to 187]

ADVERSE EVENTS:
Time Frame: 72 hours post-op
Arm/Group | Non-opiod Pain Relief
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03714919/Prot_001.pdf